CLINICAL TRIAL: NCT01333852
Title: Randomized Phase II Study of Paclitaxel Plus Metformin or Placebo for the Treatment of Platinum-refractory, Recurrent or Metastatic Head and Neck Neoplasms
Brief Title: Metformin Plus Paclitaxel for Metastatic or Recurrent Head and Neck Cancer
Acronym: METTAX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Lucas Vieira dos Santos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); University of Campinas, Brazil (Other)
Responsible Party: Sponsor-Investigator, Lucas Vieira dos Santos, Dr, Barretos Cancer Hospital
Organization: Barretos Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: METTAX200901
Record Dates: First submitted 2011-04-05; First posted 2011-04-12 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Head and Neck Neoplasms; Squamous Cell Carcinoma
Keywords: head and neck cancer; paclitaxel; metformin; squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel, placebo (Active Comparator): Paclitaxel 175mg/m² q21d until disease progression, unacceptable toxicity or consent withdrawal
  Interventions: Drug: paclitaxel 175mg/m² q21d; Drug: placebo
- Paclitaxel plus metformin (Experimental): Paclitaxel 175mg/m² q21d + metformin up to 2500mg/d until disease progression, prohibitive toxicity or consent withdrawal
  Interventions: Drug: metformin up to 2500mg/d; Drug: paclitaxel 175mg/m² q21d

INTERVENTIONS:
Drug: metformin up to 2500mg/d — metformin up to 2500mg/d
  Other Names: Glifage
  Arms: Paclitaxel plus metformin
Drug: paclitaxel 175mg/m² q21d — paclitaxel 175mg/m² q21d
  Other Names: taxol
Drug: placebo — placebo
  Arms: Paclitaxel, placebo

SUMMARY:
Metformin plus paclitaxel for recurrent or metastatic head and neck cancer: a randomized phase II trial

DETAILED DESCRIPTION:
METTAX is a phase II randomized trial that aim to evaluate the addition of metformin to paclitaxel in patients that failed to curative-intent treatment for Head-and neck neoplasms.

Patients eligible for this protocol will be randomized to paclitaxel 175mg/m2 plus metformin or placebo until disease progression or unacceptable toxicity. The primary end-point is disease control (complete response, partial response or stable disease, according to RECIST 1.1) in the 12th week. Secondary end-points are PFS, OS, response rate and safety. Molecular markers in samples collected before and under treatment will be tested for correlation with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Biopsy-proven head and neck squamous cell carcinoma
* Ineligibility for curative intent therapy, e.g., surgery or radiation therapy
* recurrent or stage IV disease
* previous failure to platinum-based chemotherapy
* measurable disease according to RECIST v1.1
* PS ECOG 0-2

Exclusion Criteria:

* known hypersensitivity to metformin or paclitaxel
* SNC metastasis
* Acute or chronic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-02; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Disease control at week 12 | 12th week
  Number of subjects at week 12 with complete response, partial response or stable disease, over the total number of subjects, for each arm. Disease control means complete response, partial response or stable disease, according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival | 6mo after the last patient recruited
  We will measure the number of subjects without progressive disease (complete response, partial response or stable disease) 6mo after the start of therapy, also after 1 and 2 years from the start of therapy. PFS will also be analysed with log-rank test, and reported as HR with respective 95% CI and p value, and median PFS will be estimated with kaplan-meyer method. All calculations will be performed 6 months after the last patient recruited. Also, the survival rate at year one and two will be calculated.
Overall Survival (subjects without death (any cause)) | 6mo after the last enrolled patient
  We will measure the number of subjects without death (any cause) 6mo after the start of therapy, and also after 1 and 2 years from the start of therapy. OS will also be analysed with log-rank test, and reported as HR with respective 95% CI and p value, and median OS will be estimated with kaplan-meyer method. All calculations will be performed 6 months after the last patient recruited. Also, the survival rate at year one and two will be calculated.
Number of patients with Grade 3-5 Adverse Events in each arm, for each category of AE | 6 mo after the last enrolled patients
  Safety and tolerability will be assessed using NCI CTCAE v3. The number of patients in each arm experiencing grade 3-5 AE (for each AE) over the total number of subjects will be measured, and the proportion of patients experiencing AE in each arm will be compared using uncorrected chi-sq test. AE will be recorded in baseline and in each visit, and the worst grade AE will be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas V dos Santos, MD, Principal Investigator — HCB; Jose BC Carvalheira, MD, PhD, Study Chair — University of Campinas, Brazil; Andre L. Carvalho, MD, PhD, Study Director — HCB
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil